CLINICAL TRIAL: NCT02775422
Title: Comparison of Serological Tests for the Varicella-zoster Virus and Correlation With the Memory of the Infection or Vaccination
Brief Title: Comparison of Serological Test s for the Virus Chicken Pox Virus (VZV) and Correlation With the Patient's Memory of the Infection or Vaccination
Acronym: VARI-IMM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low inclusion rate.
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014/08; 2014-A00707-40 (Other: ANSM)
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2019-08

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant women (Experimental): Pregnant women
  Interventions: Biological: Serological Test s for the Virus Chicken Pox Virus

INTERVENTIONS:
Biological: Serological Test s for the Virus Chicken Pox Virus

SUMMARY:
Comparison of the sensibility and specificity of 3 different serological tests and evaluation of chicken pox immunity in pregnant women.

Secondary goals :

* Correlation memory / Immunity;
* Prevalence of VZV immunity in pregnant women;
* Evaluation of cellular and humoral immunity in cases with discrepancy between tests or between test and memory;
* Evaluation of acceptability of vaccination in the post partum period in non immune patients.

Methods Not randomized prospective study,

Number of patients : 400 Duration : 36 months Inclusion criteria : pregnant women >18years old, agree to participate (written consent) Exclusion criteria: auto immune disease, HIV +, grafted patients

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged over 18
* Affiliated to a social protection scheme or women benefiting from such a regime
* Women who gived a writing consent

Exclusion Criteria:

* Women with a maternal disease: autoimmune disease (systemic lupus erythematosus, antiphospholipid syndrome, insulin dependent diabetes, autoimmune thyroiditis ..), it takes an immunosuppressive treatment or not.
* HIV-positive women
* Garfted women whatever organ

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2020-07-26 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
Rate sensitivity and specificity in negative and dubious zone for the assessment of the serology of anti VZV immunity | 35 weeks

SECONDARY OUTCOMES:
frequency of immunity detecting depending on whether the patient remember having varicella, have been in contact with next of kin with varicella or been vaccinated against varicella or not | up to 35 weeks
Percentage of women accepting the vaccination in case of negative history | day during the first visit

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Picone, MD, Principal Investigator — Service Gynécologie Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LAFORET EG, LYNCH CL Jr. Multiple congenital defects following maternal varicella; report of a case. N Engl J Med. 1947 Apr 10;236(15):534-7. doi: 10.1056/NEJM194704102361504. No abstract available. PMID 20293114
- [Background] Alkalay AL, Pomerance JJ, Rimoin DL. Fetal varicella syndrome. J Pediatr. 1987 Sep;111(3):320-3. doi: 10.1016/s0022-3476(87)80447-x. No abstract available. PMID 3625399
- [Background] SAUERBREI A. Fetales varizellen syndrom. Monatsschr kinderheiledkd 2003;151:209-213.
- [Background] Miller E, Cradock-Watson JE, Ridehalgh MK. Outcome in newborn babies given anti-varicella-zoster immunoglobulin after perinatal maternal infection with varicella-zoster virus. Lancet. 1989 Aug 12;2(8659):371-3. doi: 10.1016/s0140-6736(89)90547-3. PMID 2569560
- [Background] ENDERS G. Varicella and herpes zoster in pregnancy and the newborn. . Varicella-zoster virus and clinical management. Arvin AM and Gershon AA, eds; UK: Cambridge University Press 2000:317-347.
- [Background] MIRLESSE V. Varicelle et grossesse. Les virus transmissibles de la mère à l'enfant. Denis F. Ed John Libey Eurotext, In Montrouge 1999:252-269.
- [Background] Khoshnood B, Debruyne M, Lancon F, Emery C, Fagnani F, Durand I, Floret D. Seroprevalence of varicella in the French population. Pediatr Infect Dis J. 2006 Jan;25(1):41-4. doi: 10.1097/01.inf.0000195636.43584.bb. PMID 16395101
- [Background] Wu MF, Yang YW, Lin WY, Chang CY, Soon MS, Liu CE. Varicella zoster virus infection among healthcare workers in Taiwan: seroprevalence and predictive value of history of varicella infection. J Hosp Infect. 2012 Feb;80(2):162-7. doi: 10.1016/j.jhin.2011.11.011. Epub 2011 Dec 19. PMID 22188630
- [Background] Vandersmissen G, Moens G, Vranckx R, de Schryver A, Jacques P. Occupational risk of infection by varicella zoster virus in Belgian healthcare workers: a seroprevalence study. Occup Environ Med. 2000 Sep;57(9):621-6. doi: 10.1136/oem.57.9.621. PMID 10935943
- [Background] Alp E, Cevahir F, Gokahmetoglu S, Demiraslan H, Doganay M. Prevaccination screening of health-care workers for immunity to measles, rubella, mumps, and varicella in a developing country: What do we save? J Infect Public Health. 2012 Apr;5(2):127-32. doi: 10.1016/j.jiph.2011.11.003. Epub 2012 Jan 18. PMID 22541258
- [Background] Almuneef M, Memish ZA, Abbas ME, Balkhy HH. Screening healthcare workers for varicella-zoster virus: can we trust the history? Infect Control Hosp Epidemiol. 2004 Jul;25(7):595-8. doi: 10.1086/502445. PMID 15301033
- [Background] Saadatian-Elahi M, Mekki Y, Del Signore C, Lina B, Derrough T, Caulin E, Thierry J, Vanhems P. Seroprevalence of varicella antibodies among pregnant women in Lyon-France. Eur J Epidemiol. 2007;22(6):405-9. doi: 10.1007/s10654-007-9136-z. Epub 2007 May 30. PMID 17534728
- [Background] Reignier F, Romano L, Thiry N, Beutels P, Van Damme P, Fau C, Gaspard C, Mamoux V, Zanetti A, Floret D. [Varicella-zoster virus seroprevalence in nursery and day-care workers in Lyon (France)]. Med Mal Infect. 2005 Apr;35(4):192-6. doi: 10.1016/j.medmal.2005.01.007. French. PMID 15914287
- [Background] Dashraath P, Ong ES, Lee VJ. Seroepidemiology of varicella and the reliability of a self-reported history of varicella infection in Singapore military recruits. Ann Acad Med Singap. 2007 Aug;36(8):636-41. PMID 17767333
- [Background] Fung LW, Lao TT, Suen SS, Chan OK, Lau TK, Ngai KL, Chan PK, Leung TY. Seroprevalence of varicella zoster virus among pregnant women in Hong Kong: comparison with self-reported history. Vaccine. 2011 Oct 26;29(46):8186-8. doi: 10.1016/j.vaccine.2011.08.090. Epub 2011 Sep 10. PMID 21911021
- [Background] Pourahmad M, Davami MH, Jahromi AR. Evaluation of anti-varicella antibody in young women before their marriage: A sero-epidemiologic study in Iran. J Clin Virol. 2010 Aug;48(4):260-3. doi: 10.1016/j.jcv.2010.04.015. Epub 2010 Jun 9. PMID 20538515
- [Background] Perella D, Fiks AG, Jumaan A, Robinson D, Gargiullo P, Pletcher J, Forke CM, Schmid DS, Renwick M, Mankodi F, Watson B, Spain CV. Validity of reported varicella history as a marker for varicella zoster virus immunity among unvaccinated children, adolescents, and young adults in the post-vaccine licensure era. Pediatrics. 2009 May;123(5):e820-8. doi: 10.1542/peds.2008-3310. PMID 19403475
- [Background] Koturoglu G, Kurugol Z, Turkoglu E. Seroepidemiology of varicella-zoster virus and reliability of varicella history in Turkish children, adolescents and adults. Paediatr Perinat Epidemiol. 2011 Jul;25(4):388-93. doi: 10.1111/j.1365-3016.2010.01180.x. Epub 2011 Apr 3. PMID 21649681
- [Background] Enders G, Miller E, Cradock-Watson J, Bolley I, Ridehalgh M. Consequences of varicella and herpes zoster in pregnancy: prospective study of 1739 cases. Lancet. 1994 Jun 18;343(8912):1548-51. doi: 10.1016/s0140-6736(94)92943-2. PMID 7802767
- [Background] Breuer J, Schmid DS, Gershon AA. Use and limitations of varicella-zoster virus-specific serological testing to evaluate breakthrough disease in vaccinees and to screen for susceptibility to varicella. J Infect Dis. 2008 Mar 1;197 Suppl 2:S147-51. doi: 10.1086/529448. PMID 18419389
- [Background] Maple PA, Rathod P, Smit E, Gray J, Brown D, Boxall EH. Comparison of the performance of the LIAISON VZV-IgG and VIDAS automated enzyme linked fluorescent immunoassays with reference to a VZV-IgG time-resolved fluorescence immunoassay and implications of choice of cut-off for LIAISON assay. J Clin Virol. 2009 Jan;44(1):9-14. doi: 10.1016/j.jcv.2008.08.012. Epub 2008 Sep 27. PMID 18823815
- [Background] Sauerbrei A, Schafler A, Hofmann J, Schacke M, Gruhn B, Wutzler P. Evaluation of three commercial varicella-zoster virus IgG enzyme-linked immunosorbent assays in comparison to the fluorescent-antibody-to-membrane-antigen test. Clin Vaccine Immunol. 2012 Aug;19(8):1261-8. doi: 10.1128/CVI.00183-12. Epub 2012 Jun 20. PMID 22718131
- [Background] Tischer A, Gassner M, Richard JL, Suter-Riniker F, Mankertz A, Heininger U. Vaccinated students with negative enzyme immunoassay results show positive measles virus-specific antibody levels by immunofluorescence and plaque neutralisation tests. J Clin Virol. 2007 Mar;38(3):204-9. doi: 10.1016/j.jcv.2006.12.017. Epub 2007 Feb 7. PMID 17289430
- [Background] Mancuso JD, Krauss MR, Audet S, Beeler JA. ELISA underestimates measles antibody seroprevalence in US military recruits. Vaccine. 2008 Sep 8;26(38):4877-8. doi: 10.1016/j.vaccine.2008.06.028. Epub 2008 Jun 27. PMID 18586062
- [Background] Seward JF, Watson BM, Peterson CL, Mascola L, Pelosi JW, Zhang JX, Maupin TJ, Goldman GS, Tabony LJ, Brodovicz KG, Jumaan AO, Wharton M. Varicella disease after introduction of varicella vaccine in the United States, 1995-2000. JAMA. 2002 Feb 6;287(5):606-11. doi: 10.1001/jama.287.5.606. PMID 11829699